CLINICAL TRIAL: NCT03066791
Title: Pilot Study on the Effects of Oral Curcumin and Turmeric on Sebum Production
Brief Title: Turmeric and Curcumin on Sebum Production
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 850932
Record Dates: First submitted 2016-11-01; First posted 2017-02-28 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Inflammation; Skin
MeSH Terms: conditions — Dermatitis | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Turmeric group (Active Comparator): Turmeric Tablets:
  Each tablet contains 1,000 mg of Turmeric (Curcuma Longa) per tablet. Dose: subjects will take 6 tablets per day, with a total daily dose of 6,000 mg.
  Supplied by Sabinsa Corporation
  Interventions: Dietary Supplement: Turmeric tablets
- Curcumin Group (Active Comparator): Curcumin and Bioperine tablets:
  Each tablet contains 1,000mg Curcumin + 1.25mg black pepper. Dose: subjects will take 6 tablets per day, with a total dose of 6,000mg curcumin.
  Supplied by Sabinsa corporation
  Interventions: Dietary Supplement: Curcumin and Bioperine tablets
- Placebo Group (Placebo Comparator): Placebo tablets made to look like the turmeric and curcumin tablets
  Each placebo tablet will contain: microcrystalline cellulose, dicalcium phosphate, PVPK30, sodium starch glycolate, magnesium stearate, OpaDry orange coating.
  Dose: subjects in this group will take 6 placebo tablets per day
  Interventions: Dietary Supplement: Placebo tablets

INTERVENTIONS:
Dietary Supplement: Turmeric tablets
  Arms: Turmeric group
Dietary Supplement: Curcumin and Bioperine tablets
  Arms: Curcumin Group
Dietary Supplement: Placebo tablets
  Arms: Placebo Group

SUMMARY:
A noticeably increasing number of patients are asking for naturally based extracts and ingredients as supplementary dermatologic remedies. Patients are seeking natural and cost-effective skin care alternatives in place of prescription medications and procedures. Our study will evaluate the effects of oral curcumin and turmeric on sebum production in healthy subjects.

DETAILED DESCRIPTION:
Turmeric extracts and curcumin have been shown to be safe, even at high doses without significant side-effects. Previous clinical studies in other inflammatory skin diseases have shown that a dosage of curcumin at 6,000 mg daily was effective while lower doses were not. In a human phase I clinical trial examining the effects of high dose curcumin in preventing premalignant lesions, even curcumin doses as high as 8,000 mg/day resulted in no toxic effects after 3 months. This study will involve participant ingestion of 6,000 mg/day of turmeric or curcumin to assess how this affects their sebum production.

The investigators will also be collecting stool from the study subjects, and examining how the curcumin and turmeric may modulate their gut microbiome. The investigators will specifically be looking to see if curcumin or turmeric have any changes on the gut flora towards bacteria that produce more short chain fatty acids. Certain bacteria that make up the microbiome produce short chain fatty acids, such as butyrate and propionate, which have demonstrated anti-inflammatory properties. Thus, it would be interesting to see if turmeric or curcumin exert any of its anti-inflammatory effects via modulation of the microbiome.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 50 years of age, and
2. Subject must be able to read and comprehend study procedures and consent forms.

Exclusion Criteria:

1. Subject should be generally healthy and have no smoking history in the past one year, and must have no history of diabetes, metabolic syndrome, known cardiovascular disease, malignancy, kidney disease, or chronic steroid use.
2. Those who used topical medications in the past two weeks or systemic antibiotics or oral probiotics within one month of starting the study.
3. Subjects who are postmenopausal
4. Those who are pregnant or breastfeeding.
5. Those that are prisoners or cognitively impaired.
6. Those who have a known allergy to black pepper should not participate in this clinical trial, since one of the treatments consists of tablets containing a small amount (1.25mg/tablet) of black pepper.
7. Those that are taking angiotensin converting enzyme inhibitor medications or angiotensin receptor blocker medications for any reason.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
Sebum production | 8 weeks
  Sebutapes will be used to measure sebum production at each visit. The sebutapes will then be collected and analyzed for fatty acids and lipid production.

SECONDARY OUTCOMES:
Change from Baseline in Sebum profile, such as inflammatory markers at 8 weeks | 8 weeks
Change in stool microbiome diversity (optional collections for subjects) from baseline at 8 weeks | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Raja K Sivamani, M.D., Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Dermatology Clinical Trials Unit, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thangapazham RL, Sharma A, Maheshwari RK. Beneficial role of curcumin in skin diseases. Adv Exp Med Biol. 2007;595:343-57. doi: 10.1007/978-0-387-46401-5_15. PMID 17569219
- [Background] Chainani-Wu N. Safety and anti-inflammatory activity of curcumin: a component of tumeric (Curcuma longa). J Altern Complement Med. 2003 Feb;9(1):161-8. doi: 10.1089/107555303321223035. PMID 12676044